CLINICAL TRIAL: NCT02630199
Title: Phase I, Open-Label Study of AZD6738, DNA Damage Repair/Novel Anti-cancer Agent, in Combination With Paclitaxel, in Refractory Cancer
Brief Title: Study of AZD6738, DNA Damage Repair/Novel Anti-cancer Agent, in Combination With Paclitaxel, in Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD,Division of hematology-oncology,Department of medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-10-038
Record Dates: First submitted 2015-12-06; First posted 2015-12-15 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Refractory Cancer
MeSH Terms: conditions — Neoplasms | interventions — ceralasertib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD6738 + paclitaxel (Experimental): The PART A will be in combination with paclitaxel; the starting dose of 40 mg AZD6738 OD will be escalated to reach a maximum tolerated dose in patients with advanced solid malignancies, as defined by dose-limiting toxicity. The PART B will be an independent parallel PK expansion cohort with cycle 0 of AZD6738 on D1, D8~D21 monotherapy followed by combination therapy with weekly paclitaxel from cycle 1.
  Interventions: Drug: AZD6738; Drug: Paclitaxel

INTERVENTIONS:
Drug: AZD6738 — The starting dose of 40 mg AZD6738 OD will be escalated to reach a maximum tolerated dose in patients with advanced solid malignancies, as defined by dose-limiting toxicity.
Drug: Paclitaxel — Paclitaxel 80mg/m2 on days 1,8, and 15 every 4 weeks

SUMMARY:
This study is a single center open label phase I study of AZD6738, DNA damage repair/novel cancer agent, in combination with paclitaxel in metastatic cancer patients who have failed standard chemotherapy.

AZD6738 is an orally dosed selective and potent inhibitor of Ataxia Telangiectasis and Rad3 Related (ATR) kinase with good selectivity against other Pi3 kinase family members.

ATR is a serine/threonine protein kinase and member of the phosphatidylinositol 3-kinase related kinase (PIKK) family. During normal replication, ATR is recruited at stalled replication forks which can progress to double strand breaks if left unrepaired. ATR is also recruited to single strand DNA coated with Replication Protein A (RPA) following single strand DNA damage or the resection of double strand breaks. Recruitment and activation of ATR leads to cell cycle arrest in the S phase while the DNA is repaired and the stalled replication fork resolved, or nuclear fragmentation and entry into programmed cell death (apoptosis).

In the clinic ATR inhibitors are expected to cause growth inhibition in tumour cells dependent upon ATR for DNA repair e.g. ATM-deficient tumours. In addition to monotherapy activity, ATR inhibitors are also predicted to potentiate the activity of cytotoxic DNA damaging agents and radiotherapy (through inhibition of ATR-dependent DNA repair processes) when used in combination. While significant enhancement of anti-tumour activity may be achieved, data with AZD6738 suggest the potential need to reduce the ATR inhibitor dose and intensity (relative to monotherapy dose) and introduce dosing breaks to allow normal tissue recovery when used in combination with systemic DNA damaging chemotherapy agents, in order to maintain tolerable therapeutic margins.

The mechanism of action of AZD6738 suggests the potential to combine it with a number of anti-cancer treatments, resulting in either synergistic or additive activity. This study is evaluating the safety, tolerability, pharmacokinetics and anti-tumour activity of AZD6738 at increasing doses, in combination with paclitaxel as one of standard salvage regimen in patients with advanced cancer.

The study will consist of two parts, each evaluating the safety and tolerability of a specific combination agent, paclitaxel with different drug schedules. An oral formulation of AZD6738 will be used.

The PART A will be in combination with paclitaxel; the starting dose of 40 mg AZD6738 OD will be escalated to reach a maximum tolerated dose in patients with advanced solid malignancies, as defined by dose-limiting toxicity. The PART B will be an independent parallel PK expansion cohort with cycle 0 of AZD6738 on D1, D8~D21 monotherapy followed by combination therapy with weekly paclitaxel from cycle 1. Investigators will modify to recruit the minimum or maximum number of patients depending on data generated from other studies using AZD6738.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be > 19 years of age.
3. Refractory cancer patients who have failed to standard of care chemotherapy.
4. Provision of tumor sample (from either a resection or biopsy): however this criteria is optional for this study (i.e. if no biopsy sample available, not an exclusion criteria).
5. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations. Especially, patients must fast (water to drink only) from at least 2 hours prior to taking a dose to at least 1 hour post-dose for all doses.
6. ECOG performance status 0-1
7. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
8. At least one measurable lesion that can be accurately assessed by imaging at baseline and following up visits.
9. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment.

   Patients of child-bearing potential should be using adequate contraceptive measures (two forms of highly reliable methods) should not be breast feeding and must have a negative pregnancy test prior to start of dosing.or Patients must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:
10. Male patients must be willing to use barrier contraception for the duration of the study and:

    * for one week after the last dose of study drug if the sexual partner is not of child bearing potential
    * for 6 months after last dose of study drug and in combination with a highly reliable contraceptive method for sexual partners of child-bearing potential
11. Male patients must be willing to not donate sperm for the duration of study or up to 6 months after the last dose of study drug.

Exclusion Criteria:

1. More than four prior chemotherapy regimens (excluding adjuvant chemotherapy) for cancer treatment
2. Any previous treatment with ATR inhibitors (small molecules)
3. Any previous treatment with paclitaxel (docetaxel is allowed if in physician's discretion, the tumor is not absolutely refractory to taxane)
4. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
5. Patients unable to swallow orally administered medication.
6. Treatment with any investigational product during the last 14 days before the enrollment (or a longer period depending on the defined characteristics of the agents used).
7. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
8. - Concomitant use of known potent CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir.

   - Receiving, or having received, concomitant medications, herbal supplements and/or foods that significantly modulate CYP3A4 or Pgp activity (wash out periods of two weeks, but three weeks for St. John's Wort). Note these include common azole antifungals, macrolide antibiotics and other medications listed in Appendix I.
9. With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy.
10. Intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
11. Resting ECG with measurable QTcF > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
12. Patients with cardiac problem as follows: uncontrolled hypertension or hypotension (BP ≥150/95 mmHg despite medical therapy, BP <100/60 mmHg or orthostatic hypotension fall in BP >20 mmHg) Left ventricular ejection fraction <55% measured by echocardiography, Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest , Symptomatic heart failure (NYHA grade II-IV), Prior or current cardiomyopathy, Severe valvular heart disease, Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy), Acute coronary syndrome within 6 months prior to starting treatment
13. Female patients who are breast-feeding or child-bearing
14. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
15. A diagnosis of ataxia telangiectasia
16. Inadequate bone marrow and impaired hepatic or renal function as demonstrated by any of the following laboratory values:

    * Haemoglobin < 9.0 g/dL (transfusion allowed)
    * Absolute neutrophil count (ANC) <1.5 x 109/L
    * White blood cells (WBC) ≤ 3 x 109/L
    * Platelet count < 100 x 109/L (transfusion allowed)
    * Albumin < 33g/L
    * Total bilirubin < 1.5 x institutional upper limit of normal (ULN)
    * AST (SGOT)/ALT (SGPT) > 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be > 5x ULN
    * Serum creatinine > 1.5 x institutional ULN
    * Glomerular filtration rate (GFR) < 45 mL/min, as assessed using the standard methodology at the investigating centre (i.e. cockcroft-Gault, MDRD or CKD-EPI formulae, EDTA clearance or 24 h urine collection)
    * Haematuria: +++ on microscopy or dipstick
    * INR ≥ 1.5 or other evidence of impaired hepatic synthesis function
17. Previous allogenic bone marrow transplant
18. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Number of participants With Abnormal Laboratory Values and/or Adverse Events to assess Safety and tolerability of AZD6738. | From baseline until 28 days after discontinuation of study treatment, assessed up to 12 months
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 to determine maximal tolerate dose (MTD) of AZD6738. | Up to 6 months

SECONDARY OUTCOMES:
Objective Response rate | expected average of 1 years
Overall survival (OS) | expected average of 1 years
progression-free survival (PFS) | expected average of 1 years
Area under the plasma concentration versus time curve (AUC) after single and multiple dose | Day 0 and Day 1
Peak Plasma Concentration (Cmax) | Day 0 and Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Korea, South Korea